CLINICAL TRIAL: NCT02859194
Title: The Effect of Lt to Rt Shunt Using Veno-veno-arterial Extracorporeal Membrane Oxygenation (ECMO) on Coronary Oxygenation in Lung Transplantation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0124
Record Dates: First submitted 2016-07-21; First posted 2016-08-08 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Interstitial Pulmonary Fibrosis ARDS; COPD (Chronic Obstructive Pulmonary Disease); Bronchiectasis; Lymphangioleiomyomatosis; Primary Pulmonary Hypertension; ARDS (Acute Respiratory Distress Syndrome)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis; Lymphangioleiomyomatosis; Familial Primary Pulmonary Hypertension; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Veno-veno-arterial ECMO group (Experimental)
  Interventions: Procedure: Veno-veno-arterial ECMO

INTERVENTIONS:
Procedure: Veno-veno-arterial ECMO

SUMMARY:
ECMO(Extracorporeal membrane oxygenation) is being essential for cardiopulmonary failure patients. There are two types of ECMO, which is veno-veno (V-V) that can be used in respiratory failure patients and veno-arterial (V-A) that can be used in cardiac failure patients. V-A ECMO can also be used during lung transplantation, substitution of cardiopulmonary bypass, which can show sufficient performance during operation and better postoperative outcome. However, regarding V-A ECMO circulating from femoral vein to femoral artery, there is a pro blem of differential hypoxia which might influence coronary artery and head vessels. In this prospective study, the investigators are planning to put another ECMO catheter into internal jugular vein which takes a role of left to right shunt, to mitigate the hypoxia of coronary artery.

ELIGIBILITY:
Inclusion Criteria:

1. scheduled for double lung transplantation

Exclusion Criteria:

1. patients who have history of coronary artery occlusive disease
2. patients with arrhythmia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
arterial blood oxygen partial pressure (PaO2) | 5 min after jugular catheter flow 0ml/min
arterial blood oxygen partial pressure (PaO2) | 5 min after jugular catheter flow 500 ml/min
arterial blood oxygen partial pressure (PaO2) | 5 min after jugular catheter flow 1,000ml/min
arterial blood oxygen partial pressure (PaO2) | 5 min after jugular catheter flow 1,500ml/min

SECONDARY OUTCOMES:
venous blood oxygen partial pressure (PvO2) | 5 min after jugular catheter flow 0ml/min
venous blood oxygen partial pressure (PvO2) | 5 min after jugular catheter flow 500 ml/min
venous blood oxygen partial pressure (PvO2) | 5 min after jugular catheter flow 1,000ml/min
venous blood oxygen partial pressure (PvO2) | 5 min after jugular catheter flow 1,500ml/min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No